CLINICAL TRIAL: NCT06983379
Title: Oxidative Stress and Vitamin D Levels in Autism Spectrum Disorders: An Original Clinical Investigation
Brief Title: Oxidative Stress and Vitamin D Levels in Autism Spectrum Disorders
Status: Completed | Type: Observational
Sponsor: Mardin Artuklu University (Other)
Collaborators: Alanya Alaaddin Keykubat University (Other)
Responsible Party: Principal Investigator, Hasan Basri Savas, Associate Professor, Mardin Artuklu University
Other Study IDs: 10354421-2019/5
Record Dates: First submitted 2025-05-05; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Autism Spectrum Disorders
Keywords: oxidative stress; Vitamin D; Autism Spectrum Disorders
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Autism spectrum disorders: 38 individuals with autism spectrum disorders
- Control: 30 healthy individuals

SUMMARY:
Oxidative Stress and Vitamin D Levels in Autism Spectrum Disorders

DETAILED DESCRIPTION:
Introduction:

The etiology of Autism Spectrum Disorder (ASD) is thought to be complex. Increasing evidence in the literature shows that oxidative stress plays a role in the development and prognosis of autism. In our study, investigators aimed to investigate whether thiol disulfide balance, which is a new marker of oxidative stress, is different from that in normal children with autism spectrum disorder.

Methods A total of 68 children, 38 with autism spectrum disorder and 30 healthy controls, were included in the study. Dynamic thiol balance, total oxidant status, total antioxidant status, ischemia-modified albumin, paraoxonase 1, and arylesterase activities were measured using colorimetric methods. Routine biochemical parameters were obtained from their files and evaluated.

ELIGIBILITY:
Control group inclusion criteria:

* Healthy children who applied to the pediatric clinic for routine examination

Control group exclusion criteria:

* Children who have any chronic medical diseases or psychiatric disorders
* Children who have a family history of chronic medical diseases or psychiatric disorders

Autism spectrum disorder group inclusion criteria:

* Children with autism spectrum disorder (Diagnosis based on the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, Text Revision (DSM-5-TR))

Autism spectrum disorder group exclusion criteria:

* Children who have a family history of chronic medical diseases or psychiatric disorders

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study included children who visited the Child and Adolescent Psychiatry and Adolescent Pediatric Gastroenterology outpatient clinics.
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2020-01-03 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Oxidative stress markers | From January 2020 to Jun 2021
  Total antioxidant status (μmol Trolox equivalent/ L)
Oxidative stress markers | From January 2020 to Jun 2021
  Total oxidant status (μmol H2O2 equivalent/L)
Oxidative stress markers | From January 2020 to Jun 2021
  Paraoxonase (U/L)
Oxidative stress markers | From January 2020 to Jun 2021
  Arylesterase (Ku/l)
Oxidative stress markers | From January 2020 to Jun 2021
  Total thiol (µmol / L)
Oxidative stress markers | From January 2020 to Jun 2021
  Native thiol (µmol / L) / alb (g / l)
Oxidative stress markers | From January 2020 to Jun 2021
  Disulfide (-S-S-) (µmol / L) / alb (g/l)
Oxidative stress markers | From January 2020 to Jun 2021
  Ischemia-modified albumin (u/L)
Oxidative stress markers | From January 2020 to Jun 2021
  Oxidative stress index (arbitrary unit)

CONTACTS AND LOCATIONS:
Locations (1):
- Alanya Training and Research Hospital, Antalya, Turkey (Türkiye)